CLINICAL TRIAL: NCT03125031
Title: Comparison of Noninvasive Hemoglobin Disposable Sensors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TR26947-TP16847A
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Results first posted 2017-06-06 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group- Sensor 1 (Experimental): All subjects are enrolled into the test group and receive the Rainbow adhesive adult/pediatric sensors.
  Interventions: Device: Rainbow adhesive adult/pediatric sensor
- Group- Sensor 2 (Experimental): All subjects are enrolled into the test group and receive the Rainbow adhesive adult/neonatal sensors.
  Interventions: Device: Rainbow adhesive adult/neonatal sensor

INTERVENTIONS:
Device: Rainbow adhesive adult/pediatric sensor
  Arms: Group- Sensor 1
Device: Rainbow adhesive adult/neonatal sensor
  Arms: Group- Sensor 2

SUMMARY:
In this study, the concentration of hemoglobin within the subject's blood will be reduced in a controlled manner by administering fluids intravenously. The accuracy of two noninvasive hemoglobin sensors will be assessed by comparison to hemoglobin measurements from a laboratory analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18-40 years of age
* Weight of at least 110 lbs and less than 250 lbs for subjects under 6 feet tall.
* Physical status of ASA I of II
* Able to read and communicate in English
* Has signed written informed consent
* Female, non pregnant.

Exclusion Criteria:

* Age less than 18 yrs and greater than 40 years
* If the Warming and cooling subjects have open cuts of skin abrasions on their extremities they will be excluded because alcohol spray may be painful.
* Weight of less than 110 lbs or more than 250 lbs if the subject is less than 6 feet tall.
* Hemoglobin less than 11 g/dL
* ASA physical status of III. IV, V.
* Pregnant
* Subject has known drug or alcohol abuse
* Subject has skin abnormalities affecting the digits such as psoriasis, eczema, angioma, scar tissue, burn, fungal infection, substantial skin breakdown, nail polish or acrylic nails.
* Subject has experienced a head injury with loss of consciousness within the last year.
* Subject has known neurological and psychiatric disorder that interferes with the subjects' level of consciousness.
* Known or concurrent chronic usage of psychoactive or anticonvulsive drugs within the last 90 days, or any use in the last 7 day (i.e. tricyclic antidepressants, MAO inhibitors, Lithum, neuroleptics, anxiolytics or antipsychotics, except SSRIs).
* Subject has any medical condition which in the judgment of the investigator, renders them inappropriate for participation in this study, such as Reynauds Syndrome.
* Systolic BP >140 mmHg or Diastolic BP > 100 mmHg.
* Baseline heart rate < 50 bpm.
* Inability to tolerate sitting still or minimal movement for up to 90 minutes
* Discretion of investigator

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2014-07-10 (Actual); Primary Completion 2014-07-25 (Actual); Study Completion 2014-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Clinical Lab, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Rainbow Adhesive Adult/Pediatric Sensor: All subjects are enrolled into the test group and receive the Rainbow adhesive adult/pediatric sensors.
- Rainbow Adhesive Adult/Neonatal Sensor: All subjects are enrolled into the test group and receive the Rainbow adhesive adult/neonatal sensors.
Period: Overall Study
Arm/Group | Rainbow Adhesive Adult/Pediatric Sensor | Rainbow Adhesive Adult/Neonatal Sensor
Started | 44 | 44
Completed | 44 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Rainbow Adhesive Adult/Pediatric and Adult/Neonatal Sensors: All subjects are enrolled into the test group and receive the Rainbow adhesive sensors (adult/pediatric and adult/neonatal sensors).
Arm/Group | Rainbow Adhesive Adult/Pediatric and Adult/Neonatal Sensors
Number analyzed (Participants) | 44
Age, Customized [Count of Participants; unit: Participants]
  18-38 years | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Noninvasive Sensors by Arms Calculation
Description: Accuracy will be determined by comparing the noninvasive hemoglobin measurement of the pulse oximeter to the hemoglobin value obtained from a blood sample and calculating the arithmetic root mean square (Arms) error value. The accuracy results from both sensors will be assessed for equivalence
Time Frame: 1-5 hours
Measure: Number; unit: g/dL
Units Other Than Participants: data points
Groups:
- Group-Sensor 1: All subjects are enrolled into the test group and receive the Rainbow adhesive adult/pediatric sensors.
- Group-Sensor 2: All subjects are enrolled into the test group and receive the Rainbow adhesive adult/neonatal sensors.
Arm/Group | Group-Sensor 1 | Group-Sensor 2
Number analyzed (Participants) | 44 | 44
Number analyzed (data points) | 691 | 928
g/dL | 1.0 | 1.0

ADVERSE EVENTS:
Groups:
- Rainbow Adhesive Adult/Pediatric and Adult/Neonatal Sensors: All subjects are enrolled into the test group and receive the Rainbow adhesive sensors (adult/pediatric and adult/neonatal).
Arm/Group | Rainbow Adhesive Adult/Pediatric and Adult/Neonatal Sensors
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes